CLINICAL TRIAL: NCT03086148
Title: Effect of Low-dose Ketamine on Postoperative Depressive Symptom in Patients Undergoing Intracranial Tumor Resection (PASSION)
Brief Title: Ketamine and Postoperative Depressive Symptom-PASSION
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Associate professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-03-16
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Ketamine; Depressive Symptom; Neurosurgery; Perioperative Period
MeSH Terms: conditions — Depression | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Experimental)
  Interventions: Drug: Ketamine
- normal saline group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — Ketamine will be administrated intravenously at dural opening, with the total dose of 0.5 mg/kg and continual infusion for 40 minutes.
  Other Names: Ketamine hydrochloride
  Arms: ketamine group
Drug: Normal saline — Normal saline will be administrated intravenously at dural opening, with the total dose of 0.5 ml/kg and continual infusion for 40 minutes.
  Arms: normal saline group

SUMMARY:
Perioperative depression symptom (PDS) is one of the common mental comorbidity, and influences the clinical outcomes and prognosis. However, there is no rapid acting treatment to deal with it during the limited hospital stay. This study aims to determine whether ketamine could improve the depressive symptom of peirioperative patients. It will also examine the safety for administrating ketamine as an antidepressant intraoperatively. Meanwhile, it will show if ketamine could improve anxiety, postoperative pain or delirium. This trial also will bring great concerns on patients with perioperative mental health and explore the measures to improve their psycho-related prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Brain tumor located supratentorial area and need to receive elective craniotomy;
2. Moderate to severe depressive symptom measured by the qualified psychiatric doctors.
3. Ages between 18 and 65 years old.
4. American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

1. History of epilepsy;
2. Major depression disorder patients undergoing antidepressive therapy within 2 weeks; 3 Psychiatric illness; 4 Drug abuse; 5 History of allergy to the research drug; 6 Tumor located in the Wernick area, Broca area or the frontal pole; 7 Hyperthyroidism; 8 Patients can not cooperate with investigators on psychiatric assessments; 9 Pregnant or breast-feeding woman; 10 refuse to sign inform consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Response rate | Postoperative 3 days
  ≥50% reduction in MADRS scores from baseline value.The MADRS is a 10-item tool, with scores ranging from 0 to 60, and determining the severity of depression.

SECONDARY OUTCOMES:
The remission rate | Postoperative 3 days and discharge.
  The remission rate is defined as the absolute value of MADRS no more than 10.
Anxiety symptom | Postoperative 3 days.
  The anxious symptom is defined as HADS score no less than 11.
Postoperative delirium | Postoperative 1 day.
  Postoperative delirium will be assessed by the Confusion Assessment Method for the Intensive Care Unit Scale (CAM-ICU) at 2 hours and 1 day after surgery.
Severe pain | Postoperative 3 days.
  The incidence of severe pain within first postoperative three days, which is defined as mean and peak numerical rating scale (NRS) are higher than 5.
Postoperative 30-day quality of life reported by KPS | Postoperative 30 days
  The quality of life will be evaluated by Karnofsky performance status (KPS) at postoperative 30 days.
Psychiatric outcomes and complications | Postoperative 3 days and discharge.
  Postoperative complications include psychiatric symptoms evaluated by Brief Psychiatric Rating Scale (BPRS), manic symptoms assessed through the 11-item Young Mania Rating Scale (YMRS), and dissociative symptoms measured by the Clinician Administered Dissociative States Scale (CADSS). Moreover, postoperative complications also include aphasia, epilepsy, hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Study Chair — Department of Anesthesiology, Beijing Tiantan Hospital
Locations (1):
- Beijing TianTan Hospital, Beijing, China

REFERENCES:
- [Derived] Zhou Y, Sun W, Zhang G, Wang A, Lin S, Chan MTV, Peng Y, Wang G, Han R. Ketamine Alleviates Depressive Symptoms in Patients Undergoing Intracranial Tumor Resection: A Randomized Controlled Trial. Anesth Analg. 2021 Dec 1;133(6):1588-1597. doi: 10.1213/ANE.0000000000005752. PMID 34633992
- [Derived] Zhou Y, Peng Y, Fang J, Sun W, Zhang G, Zhen L, Wang G, Han R. Effect of low-dose ketamine on PerioperAtive depreSsive Symptoms in patients undergoing Intracranial tumOr resectioN (PASSION): study protocol for a randomized controlled trial. Trials. 2018 Aug 29;19(1):463. doi: 10.1186/s13063-018-2831-0. PMID 30157913